CLINICAL TRIAL: NCT01539447
Title: Influence of Naproxen on Heterotropic Bone Formation Following Hip Arthroscopy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Stephen Aoki, M.D., University of Utah
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 48961
Record Dates: First submitted 2012-01-12; First posted 2012-02-27 (Estimated); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Heterotopic Ossification
Keywords: Hip arthroscopy; Femoroacetabular impingement; Heterotopic ossification; Heterotopic bone formation
MeSH Terms: conditions — Ossification, Heterotopic; Femoracetabular Impingement | interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Naproxen (Active Comparator): • Group 1: Naproxen 500 mg twice daily for three weeks following surgery beginning postoperative day #1
  Interventions: Drug: Naproxen
- Placebo (Placebo Comparator): • Group 2: Placebo twice daily for three weeks following surgery beginning postoperative day #1
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Naproxen — • Group 1: Naproxen 500 mg twice daily for three weeks following surgery beginning postoperative day #1
  Arms: Naproxen
Drug: placebo — • Group 2: Placebo twice daily for three weeks following surgery beginning postoperative day #1
  Other Names: Placebo Control
  Arms: Placebo

SUMMARY:
In a brief summary the study would like to evaluate the effectiveness of Naproxen in preventing radiographically detected heterotopic ossification following hip arthroscopy for the treatment of femoroacetabular impingement.

DETAILED DESCRIPTION:
Heterotopic bone formation (HO) is a potentially serious complication of hip surgery. HO, defined as the formation of normal bone in an abnormal soft tissue location, results from alteration in the normal regulation of skeletogenesis. Although most patients remain asymptomatic despite HO development, two articles that included 10,826 patients from 37 studies suggest HO may be associated with substantial compromise of function and range of motion even at low grades.In a large pooled incidence study, HO was estimated to be 43% in 59,121 patients undergoing total hip arthroplasty, and 51% in 998 patients after acetabular trauma.

Few studies have reported on the incidence of HO following hip arthroscopy. However, HO is an increasingly reported complication of arthroscopic treatment for femoroacetabular impingement(FAI). In a comparison of complications following arthroscopic treatment of FAI in 8 case-series, ectopic ossification occurred in up to 6% of cases and accounted for 10 of the 19 reported complications. Additionally, one recent study reported an HO incidence of 33% (5 out of 15 patients) following hip arthroscopy in patients not prophylaxed with NSAID therapy. In our experience, HO occurs at a comparable or higher rate of 10% in those undergoing this procedure. The formation of ectopic ossification is triggered as a result of muscle damage during introduction of hip portals and is potentially augmented by seeding of bone shavings in the soft tissues created during burring of the femoral neck.

Prophylaxis of HO targets the biochemical mechanisms of heterotopic bone formation by: 1) Disrupting inductive signaling pathways, 2) Altering osteoprogenitor cells in target tissues, and 3) Modifying the environment conductive to formation of heteroptic bone. The two mainstays of therapy are low dose radiation treatment and non-steroidal anti-inflammatory medications (NSAIDs). The efficacies of these treatments were found to be equivalent by Burd et al in 166 randomized patients. However, NSAID therapy was shown to be considerably more cost effective with lower rates of morbidity. Large randomized studies have subsequently shown large reductions in the incidence of HO using NSAID therapy in the perioperative period. The Cochrane review of 16 randomized trials in 5000 patients found one-half to two-thirds reduction in HO with indomethacin.Even less potent NSAID therapy has been effective in reducing rates of HO. Fransen et al reported a 30% reduction in HO during the HIPAID trial comparing perioperative ibuprofen with placebo in nearly 1000 patients. The two groups had no statistical difference in functional outcome despite the higher incidence of HO in the prophylaxed group.

While NSAID therapy has been effective in reducing the incidence of HO, it is associated with potentially serious side affects. Fransen et al found 202 GI side effects in a metaanalysis of 4328 patients taking NSAIDs for HO prophylaxis.1 Of these, 138 were minor (e.g. nausea, dyspepsia, diarrhea) and 64 were major (e.g. hematemesis or melena). Overall, there was a 31% increase in the risk of GI side effects among patients taking NSAIDs. Furthermore, NSAID therapy could impair bone and/or soft tissue healing following this. These side affects could negate the benefit of NSAID therapy, especially if HO is asymptomatic in the majority of patients.

We hypothesize that NSAID prophylaxis of HO may have a role in hip arthroscopy for the treatment of femoroacetabular impingement. All NSAIDs tested, with the exception of aspirin, have resulted in significant decreases in the incidence of HO following hip surgery including less potent regimens such as ibuprofen 1200 mg/day. Naproxen offers the advantage of twice daily dosing with similar potency to ibuprofen. It is readily available and inexpensive. Furthermore, in an unpublished series of 50 patients prescribed naproxen following hip arthroscopy for FAI, we have had no cases of HO at 6 month follow up compared to a 5-10% rate in patients who received no prophylaxis. We propose testing our hypothesis that perioperative naproxen will reduce the incidence of HO following hip arthroscopy in a placebo controlled, double-blinded, randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* The patient is 18-80 years of age.
* The patient has provided written informed consent.
* The patient is scheduled for hip arthroscopy surgery for treatment of FAI
* The patient has an ASA of I, II, or III.
* The patients understands the explanation of the protocol.

Exclusion Criteria:

* The patient has history of a major GI bleeding event
* The patients has a history of renal impairment or creatinine > 1.5
* The patient has taken NSAIDs within 48 hours of surgery or in the perioperative period
* The patient has a history of heterotopic ossification following surgery
* The patient has a hypersensitivity reaction to Naproxen
* The patient is undergoing a concomitant procedure in addition to treatment of FAI

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2012-01; Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
Number of participants with documented Heterotopic Ossification (HO) in the Naproxen group vs Placebo group | 75 days after surgery
  The hypothesis is that there will be fewer instances of HO in the Naproxen group compared to the Placebo group.

SECONDARY OUTCOMES:
Number of participants with adverse events in the Naproxen group vs Placebo group. | Data outcome collected 4 weeks post operatively
  Adverse events include GI upset, GI bleed, Kidney failure, Drug reactions and Healing problems.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Aoki, M.D., Principal Investigator — University of Utah Orthopedics Center
Locations (1):
- University of Utah Orthopedics Center, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Beckmann JT, Wylie JD, Potter MQ, Maak TG, Greene TH, Aoki SK. Effect of Naproxen Prophylaxis on Heterotopic Ossification Following Hip Arthroscopy: A Double-Blind Randomized Placebo-Controlled Trial. J Bone Joint Surg Am. 2015 Dec 16;97(24):2032-7. doi: 10.2106/JBJS.N.01156. PMID 26677237